CLINICAL TRIAL: NCT04563962
Title: Contingency Management for PrEP Adherence and/or Methamphetamine UseDisorder Among MSM and TW in Los Angeles: A Pilot Feasibility Study
Brief Title: Contingency Management for PrEP Adherence and/or Methamphetamine Use
Acronym: C-MAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Jesse Clark, Associate Professor-in-Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB#19-001996
Record Dates: First submitted 2020-09-20; First posted 2020-09-25 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Methamphetamine-dependence; HIV-1-infection
Keywords: Methamphetamine; HIV; Contingency Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency Management-ART (Experimental): Contingency management intervention with incentives tied to provision of urine samples with detectable levels of Tenofovir (TFV).
  Interventions: Behavioral: Contingency Management-ART
- Contingency Management-Methamphetamine (Active Comparator): Contingency management intervention with incentives tied to provision of urine samples with no detectable levels of methamphetamine (MA).
  Interventions: Behavioral: Contingency Management-Methamphetamine

INTERVENTIONS:
Behavioral: Contingency Management-ART — Participants in this arm will participate in a Contingency Management intervention where rewards are linked with demonstrated adherence to tenofovir-based ART or PrEP.
  Arms: Contingency Management-ART
Behavioral: Contingency Management-Methamphetamine — Participants in this arm will participate in a Contingency Management intervention where rewards are linked with demonstrated abstinence from methamphetamine use.
  Arms: Contingency Management-Methamphetamine

SUMMARY:
Use of crystal methamphetamine (MA) leads to changes in sexual risk behavior, adherence to HIV prevention tools, immune response to infection, and tissue inflammation that collectively increase risk for HIV transmission among MA-using men who have sex with men (MSM), their sexual partners, and their networks. Contingency Management (CM) offers a behavioral modification tool helpful for reducing frequency of MA use, but the effects of CM on the behavioral and biological factors that promote HIV transmission in MSM networks have only been partially evaluated. The intersection of substance use, sexual risk behavior, and HIV transmission in MSM networks presents a critical problem for contemporary HIV prevention as HIV-uninfected MSM who use MA have a 16%-33% greater risk for HIV infection, while only approximately 50% of HIV-infected MA-using MSM achieve and maintain an undetectable viral load. The investigators propose to compare two different CM models to integrate substance use treatment with HIV prevention among MA-using MSM: 1) Traditional CM targeted to MA abstinence and 2) Allternative CM based on ARV adherence.

DETAILED DESCRIPTION:
Background

The intersection of substance use, sexual behavior, and HIV transmission in the social and sexual networks of crystal methamphetamine (MA)-using men who have sex with men (MSM) presents a critical public health problem. MA use increases risk for HIV acquisition and transmission in an interwoven series of behavioral, biological, and social mechanisms. Behaviorally, MA use stimulates pleasure-seeking behavior, increasing the likelihood of high-risk sexual contacts and impairing adherence to tools like condoms, pre-exposure prophylaxis (PrEP), and Treatment as Prevention (TasP). Biologically, MA affects immunologic factors associated with HIV-1 transmission, including viral replication, inflammatory cytokine production, T-cell activation, and recruitment of CD4+ T-cells to rectal mucosa. Socially, MA use negatively impacts the perceptions of interpersonal commitment and social cohesion central to community norms of HIV prevention, while elevating the incidence of untreated HIV/STIs in the population and increasing risks of exposure for sexual network contacts. Efforts to address these problems have typically prioritized either reducing MA use or controlling HIV transmission, without targeting the overlapping space between the two problems and exploring how individual-level interventions targeted to high-risk networks can transform community-scale outcomes.

Contingency Management (CM) has been shown to control MA use among habitual users. Adapting principles of behavioral economics, CM addresses the prioritization of short-term rewards and the devaluation of long-term risks commonly seen with MA use. While behavioral approaches like Cognitive Behavioral Therapy have been evaluated as strategies to manage stimulant abuse, these methods have not shown independent benefit in modifying patterns of drug use, presumably because they do not intervene in the cognitive risk-reward feedback loop that underlies stimulant abuse and that is replaced by CM incentives. Analysis of previous clinical trial data suggests that the small financial incentives provided in exchange for stimulant-free urine may substitute for the short-term feedback loops that structure the cognitive processes of habitual MA users, and serve as an essential component in CM's success.

The potential indirect effects of CM on HIV transmission have been evaluated in several studies. In conjunction with reduced MA use, MSM often report a corresponding reduction in frequency of condomless intercourse. However, efforts to implement CM as a harm reduction strategy in sexually transmitted infection (STI) clinics have been unsuccessful, leading to questions about how it can be applied to real world settings. In these contexts, incremental improvements among individual MA users are often insufficient in modifying problems like frequency of condomless intercourse, adherence to antiretroviral therapy (ART), and network-level patterns of HIV and STI transmission. The goal of the current research is to use CM as a platform to integrate HIV prevention with substance use treatment among MA-using MSM to transform population-level patterns of HIV transmission.

Specific Aims Aim 1. To assess the logistics, feasibility, and acceptability of a point-of-care urine assay to assess short-term adherence to Tenofovir (TFV)-based antiretrovirals (ARVs) or PrEP regimens among MA-using MSM. The investigators plan to enroll 10 HIV-infected and 10 HIV-uninfected MSM with recent use of MA and a tenofovir-based HIV treatment or prevention regimen. Participants will be randomly assigned to traditional CM (Arm A) or ARV-based CM (Arm B) and asked to attend monitoring visits three times per week over a 30-day period. Each visit will include urine monitoring for recent MA use and ART adherence (in both Arms). At each visit where a participant's urine either does not contain MA (Arm A) or does contain tenofovir (Arm B), they will receive a small financial incentive. Incentives will gradually increase with each successful urine test, or they will reset to zero if the participant fails the urine screen or misses a visit. Aim 1 outcomes will assess participant retention, satisfaction and acceptability of the CM format for supporting ARV adherence.

Aim 2. To collect preliminary data on the effect of ARV-based CM in promoting ARV adherence. To design an R01 trial of CM to support ARV adherence, the investigators plan to collect preliminary effect estimates for the two CM platforms in promoting: i) MA abstinence; ii) ARV adherence, and iii) Reductions in high-risk sexual behavior. Findings will be used to project sample size and refine monitoring procedures in the larger trial.

Methods Recruitment and Screening.

The investigators will recruit active MA users from community venues. Potential subjects will be recruited by a team of experienced, community-based researchers. To avoid withholding an effective CM therapy intervention from individuals trying to limit their use, for this pilot study the investigators will only enroll MSM who are not currently seeking substance use treatment. Enrollment will be limited to individuals who:

1. Identify as male or transgender;
2. Report condomless anal intercourse with a male or transgender partner in the prior 6 months;
3. Report current MA use (at least once per week) with MA present in urine at screening; and
4. Are currently taking Truvada for PrEP (if HIV-uninfected) or a Tenofovir-based ART regimen (if HIV-infected).

   Potential participants will undergo preliminary screening by the study recruiter using an IRB-approved screening script. Eligible participants will be scheduled for an Enrollment visit at the UCLA Vine Street Clinic.

   At the Enrollment visit, all participants will be asked to provide informed consent prior to the initiation of any study procedures. Upon providing consent, participants will be assessed for eligibility by a study physician and asked to provide a urine sample to test for presence of methamphetamine metabolites.

   Eligible subjects participants will be asked to complete the following Enrollment visit procedures.

   i) Behavioral Survey: All participants will be asked to complete a computer-assisted self-administered (CASI) survey assessing their demographic characteristics, substance use practices, current use of PrEP (if HIV-uninfected) or antiretroviral therapy (if HIV-infected), sexual practices, characteristics of recent partners, and social and sexual network composition.

   ii) HIV Testing: Study counselors will provide HIV risk reduction counseling using the CDC RESPECT-2 model and test for HIV with a 5th Generation HIV-1/2 Ab assay. Positive results will be confirmed by HIV-1 PCR testing for viral load quantification. Referrals to prevention and treatment services will be provided as needed.

   iii) STI Testing: Participants will undergo syphilis testing by rapid plasma reagin (RPR) with T palladium particle agglutination (TPPA) assay confirmation and serial dilution of positive titers. Participants will be asked to provide urine, rectal and pharyngeal swabs for gonorrhea and chlamydia (GC/CT) testing. Participants with an STI will receive appropriate antibiotic treatment and partner notification counseling.

   iv) Urine Toxicology Screen: Urine samples will be tested for stimulants and other drugs of abuse using a point-of-care liquid chromatography (LC) assay.

   At the Enrollment visit, participants will be randomly assigned to a CM program with incentives based either on MA abstinence or TFV adherence and with monitoring visits either twice per week or three times per week.

   b. Contingency Management Visits. Eligible participants will be counseled on CM procedures at the Enrollment visit. Participants will be asked to return to the site either two or three times per week (T-Th or M-W-F) for 4 weeks. At each visit, participants will meet with a counselor to discuss their use of PrEP/ART, MA, and sexual risk behavior. Participants will be asked to provide a urine sample for point of care testing to detect presence of: a) Methamphetamine (MA); and b) Tenofovir (TFV). Verified MA abstinence (Arm A) OR TFV use (Arm B) for the prior 3-day period will be rewarded with an escalating series of incentives.

   If a participant fails urine testing, their incentive schedule resets to the Baseline value.

   Following Enrollment, all participants will be asked to return for Contingency Management visits two or three times per week for four weeks. Each visit will include the following procedures:

   i) Behavioral Assessment: Participants will complete a brief, 12-item CASI survey assessing recent MA use, PrEP/ART adherence, and frequency of CAI with serodiscordant/unknown status partners.

   ii) Counseling: After completing the survey, study counselors will conduct a brief check-in session using motivational interviewing techniques to encourage MA abstinence, ARV adherence, and condom use.

   iii) Urine Toxicology Screening: Urine samples will be tested for presence of MA metabolites.

   iv) Tenofovir Screening: Urine samples will be tested at point-of-care for presence of Tenofovir metabolites using an experimental assay developed by Alere with Dr. Gandhi (UCSF). Similar to urine toxicology screening, this point-of-care LC assay can be performed in 15 minutes without specialized training and detects presence of both TDF and TAF metabolites indicating Tenofovir use in the prior 3-day period.

   c. Final Visit.

   At the Final visit, participants will be asked to complete the following procedures:

   i) Behavioral Assessment: Participants will be asked to complete a CASI survey similar to the enrollment instrument, with attention to changes in sexual behavior, substance use practices, and network composition.

   ii) Biological Assessment: Participants will undergo repeat testing for HIV (including viral load, if HIV-infected) and STIs, as well as urine screening for MA and Tenofovir metabolites.

   iii) Assessment of Study Procedures: Participants will be asked to complete a structured survey evaluating their satisfaction with and specific study procedures (e.g., frequency of visits, length of visits, individual counseling, incentive structures, and perceived impact on ARV adherence, MA use, and sexual risk behavior).

ELIGIBILITY:
Inclusion Criteria:

1. Identify as male or transgender female;
2. Report sexual intercourse with a male or transgender female partner in the prior 6 months;
3. Report current MA use (at least once per week) with MA present in urine at screening; and
4. Taking Truvada or Descovy for PrEP (if HIV-uninfected) or a Tenofovir-based ART regimen (if HIV-infected).

Exclusion Criteria:

Exclusion Criteria (for all study components):

1. Inability to understand the study procedures or to provide informed consent
2. Not taking a tenofovir-based regimen for HIV prevention or treatment
3. Actively seeking treatment for Methamphetamine Use Disorder (MUD)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Intervention is designed for men who have sex with men (MSM) and transgender women.
Enrollment: 20 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
PrEP/ART Adherence | 28 days
  Proportion of visits in which there are detectable levels of tenofovir in participant urine samples.
Methamphetamine Abstinence | 28 days
  Proportion of visits in which there are no detectable methamphetamine metabolites in participant urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse L Clark, MD, Principal Investigator — University of California, Los Angeles; Monica Gandhi, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCLA Vine Street Clinic, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No